CLINICAL TRIAL: NCT02887924
Title: THE EFFECT OF SUSTAINED LUNG INFLATION MANEUVER APPLIED THROUGH NASAL PRONG ON EARLY AND LATE RESPIRATORY MORBIDITIES IN PRETERM INFANTS
Brief Title: SLI MANEUVER and RESPIRATORY MORBIDITIES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12082016
Record Dates: First submitted 2016-08-15; First posted 2016-09-02 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): SLI group In this group the preterm infants will receive sustained lung inflation (SLI) via short binasal prongs in the delivery room.
  Interventions: Device: Neopuff; Fisher and Paykel, Auckland, New Zealand
- group 2 (Placebo Comparator): Preterm infants will be assisted in the delivery room without sustained lung inflation.
  Interventions: Device: Neopuff; Fisher and Paykel, Auckland, New Zealand

INTERVENTIONS:
Device: Neopuff; Fisher and Paykel, Auckland, New Zealand — Following the oral and nasal aspirates, SLI at 25 cm H2O pressure will be applied for 15 seconds by using t-piece refreshing and binasal prongs and 5-cm nCPAP at H2O pressure will be applied.
  Other Names: SUSTAINED LUNG INFLATION MANEUVER

SUMMARY:
Purpose: The investigators hypothesis is that, as compared to the only nCPAP-applied group, application of SLI maneuver followed by respiratory support with nCPAP immediately afterwards in preterm infants at high risk for RDS would reduce the need for intubation and mechanical ventilation in early period and ultimately will improve respiratory outcomes.

DETAILED DESCRIPTION:
Primary Outcome Measures:

Surfactant need, intubation and mechanical ventilation needs within the first 72 hours of life in SLI (Sustained Lung Inflation) maneuver-applied preterm infants and non-SLI-applied preterm infants.

Secondary Outcome Measures:

* Heart rate, fractional inspiratory oxygen, CPAP pressure and oxygen saturation within the first 72 hours of life in preterm infants
* Total non-invasive, invasive respiratory support time
* The presence of and the degree of BPD (Bronchopulmonary dysplasia)
* Premature morbidities such as PDA (patent ductus arteriosus), IVH (intraventricular hemorrhage), NEC (necrotizing enterocolitis), ROP (retinopathy of prematurity)
* Feeding intolerance, reaching birth weight and transition to full oral feeding time

Study Design Randomization Group 1: Group that received SLI maneuver immediately after birth followed by nCPAP.

Group 2: Group that received nCPAP after birth. Following the oral and nasal aspirates, SLI at 25 cm H2O pressure will be applied for 15 seconds by using t-piece refreshing and binasal prongs and 5-cm nCPAP at H2O pressure will be applied.

Patients will be observed for 5-10 seconds in terms of cardiorespiratory functions following SLI maneuver. If respiratory failure continues during nCPAP (such as apnea, gasping) and/or heart rate is > 60 / min but < 100 / min , SLI maneuver will be repeated at the same pressure for the same time period. If heart rate > 60 / min but <100 / min persists after the second SLI maneuver, resuscitation will be applied in line with the guidelines of American Academy of Pediatrics.

The control group of infants will receive nCPAP support at 5 cm H2O pressure and be supported in line with the guidelines of American Academy of Pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant with gestational age of 26 weeks 0 days and 29 weeks 6 days will be included.

Exclusion Criteria:

1. Presence of major congenital anomaly,
2. Patients with hydrops fetalis and pulmonary hypoplasia
3. Consent not provided or refused

Max Age: 3 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
mechanical ventilation requirement | 72 hours
  Surfactant requirement, intubation and mechanical ventilation needs within the first 72 hours of life in SLI (Sustained Lung Inflation) maneuver-applied preterm infants and non-SLI-applied preterm infants.

IPD SHARING:
Plan to Share IPD: Undecided